CLINICAL TRIAL: NCT05387590
Title: Health Care Providers Perceptions, Ratings and Motivation to Adopt/Utilize a Novel and State of the Art Physical Wellness Assessment Device (Preventiometer)
Brief Title: Health Care Provider Preventiomter Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to conduct study due to equipment not operational from study Sponsor team in Germany
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-011313
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Wellness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preventiometer Device (Other): The Preventiometer is a physical wellness tool that assesses multiple physical wellness measures in a 60 ± 15 minutes period of time. It is intended to promote population wellness by empowering individuals to act upon the information they receive about their overall health.
  Interventions: Behavioral: Preventiometer device with wellness coaching

INTERVENTIONS:
Behavioral: Preventiometer device with wellness coaching — Four wellness coaching sessions with a certified wellness coach to develop and implement your own personalized wellness plan will be included in this study.

SUMMARY:
The purpose of this study is to evaluate health care providers' perceptions, ratings and motivation to adopt a novel and state of the art physical wellness assessment device, the Preventiometer.

DETAILED DESCRIPTION:
The Preventiometer is a physical wellness tool that assesses multiple physical wellness measurements in a 60 +/- 15 minute period of time.

ELIGIBILITY:
Inclusion Criteria:

* Health care providers practicing at Mayo Clinic.
* Able to speak English and complete surveys.
* Able to read, understand and sign inform consent.

Exclusion Criteria:

* Unable to sign inform consent.
* Pregnant women. (As verbalized by participant).
* Unable to ambulate without assistance.
* Not currently involved in another formal program or research study involving wellness coaching.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Likert scale questionnaire on Preventiometer Wellness Assessment | 1 day
  Health care providers perception of the Preventiometer Wellness Device.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials